CLINICAL TRIAL: NCT05771610
Title: Sedentary Time in Individuals With Ischaemic Heart Disease and Its Association With Cardiac Function, Structure and Cardiovascular Risk Factors
Brief Title: SB and Cardiac Function and Structure in IHD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Bedfordshire (Other)
Responsible Party: Principal Investigator, Abbie C. Bell, Principal Investigator, University of Bedfordshire
Other Study IDs: SB and IHD
Record Dates: First submitted 2023-03-02; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases; Sedentary Behavior
MeSH Terms: conditions — Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Activity pattern in CVD — Only individuals who have had a cardiac event within the past twelve months upon recruitment will be included in this study.

SUMMARY:
Cardiovascular Disease (CVD) is the leading cause of mortality and morbidity globally. Following a myocardial infarction (MI), an individual is at an increased risk of a secondary event (20-50% higher risk post MI), compared to those with no prior CVD. Independent of physical activity levels, high amounts of daily sitting is a risk factor for CVD, of which sitting is typically used as an indicator for sedentary behaviour. Sedentary behaviour is defined as a waking energy expenditure of less than 1.5 METs (metabolic task equivalent) while in a seated, reclined or lying posture.

Currently, there is little knowledge regarding the prevalence of sedentary behaviour ischaemic heart disease. The aim of this study is therefore to measure activity levels of an individual following a diagnosis of ischaemic heart disease, alongside its association to cardiac function and cardiovascular risk factors. Sitting patterns and physical activity will be monitored 24 h/day during each condition using an activPAL activity monitor (PAL Technologies, Glasco, Scotland). This will measure changes in posture and level of activity by cadence.

DETAILED DESCRIPTION:
An observational, cross-sectional study design will be used. Participants can have preliminary measures taken either during a visit to the Sport and Exercise Sciences Laboratories at the University of Bedfordshire or in their own home, depending on the participant's preference. This consists of anthropometric measures (height, weight and waist circumference). Participants will then rest for 5 minutes to achieve a steady state before baseline blood pressure is taken. Baseline cardiac function measures will be measured using an echocardiogram scan, as well as an electrocardiogram (ECG) to ensure there are no electrical contraindications to the heart (including new ST depression / elevation or any arrythmias) which would make the participant unsuitable to complete the study. Mood and wellbeing measures will then be assessed using questionnaires.

Following this, participants will be asked to complete 7 full days of normal daily activity, whilst wearing an activPAL monitor on their thigh to record sitting, standing and stepping. The main data collection will take place at the participant's home, workplace or leisure setting (i.e. under free-living conditions), with social distancing in place if required at the time of data collection. Instructions will be given to help ensure that the 7-day monitoring period reflects their usual habits. The monitoring period will also be carefully decided, to ensure it does not conflict with any events that are out of the usual for the participant, such as holidays or work-based events, which would alter their usual sedentary patterns.

Data collection

Demographic data Patient demographic data will include age, gender, diagnosis and intervention. This is routinely collected within Cardiac Rehabilitation as part of their usual standard of care.

Height and weight Equipment to measure height, weight and waist circumference will include a stadiometer (Leicester Height Scale, Marsden HM-250P, Leicester, UK) to measure height in cm, a measurement tape for waist circumference and digital weighing scales (Tanita, BWB0800, Allied Weighing, UK) to measure weight in kg.

Blood pressure and heart rate Blood pressure and heart rate will be measured in an upright, seated position using an automated device (Omron M5-1 automated oscillatory device, Omron Matsusaka Co. Ltd., Matsusaka, Japan). The left arm will be used to measure blood pressure unless there is preference for the right arm due to any potential previous medical conditions. Two measures will be taken, with 5 minutes apart.

Cardiac function In a laboratory or in the participants home, the participant will be asked to undress from the waist up and lay on the medical couch in the left lateral decubitus position. Here, a scanning gel will be applied to the echocardiogram probe. This forms part of the echocardiogram system (Esoate, MyLab Omega, Italy). Parasternal and apical views will be acquired. Once these images are collected and stored, the gel will be removed from the probe and chest. All images will be stored anonymously, where participants will be given a participant ID number. All image analysis will be completed using Echopac software (GE Healthcare, Version 113, GE healthcare, Chicago, Illinois, United States). Measures taken from the echocardiogram scan will be used to calculate left ventricular structure and function.

Anxiety and Depression The Hospital Anxiety and Depression Scale will be used to assess feelings of anxiety or depression.

Measurement of sitting, standing and light physical activity Following preliminary measures, sitting, standing and stepping will be monitored 24 h/day over seven full days using an activPAL activity monitor (PAL Technologies, Glasco, Scotland). This will measure changes in posture and level of activity by cadence. The activity monitor will be attached to the skin with a waterproof dressing on the anterior right thigh. standing. The Processing PAL application will be used to process the data collected from the activPAL device. It uses a vaildated algorithm to isolate waking and sleeping time and to generate the outcome data. Participants will also be given a 7 day activity diary to record waking times, and other relevant activities to cross-validate the Processing PAL measured sleep and wake times.

ELIGIBILITY:
Inclusion Criteria:

* · Patients diagnosed with ischemic heart disease within the past 12 months (within National Audit of Cardiac Rehabilitation (NACR) outcome data). This includes post myocardial infarction (ST wave elevated MI or Non-ST wave elevated MI), post coronary artery bypass graft, post percutaneous coronary intervention.

  * Males and females
  * Aged 18 years or above.
  * Any ethnicity.

Exclusion Criteria:

* · Under 18 years of age.

  * Unable to provide valid informed consent (lack of mental capacity).
  * Not had a cardiac event diagnosed within the past 12 months.
  * Unstable coronary disease.
  * Disease or conditions with a prognosis of less than 6 months to end of life (palliative care).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ischaemic heart disease, including a myocardial infarction within the past twelve months ((NSTEMI or STEMI) confirmed by blood markers or electrophysiological changes); or angina treated with PCI or CABG.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2023-03-06 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Daily sitting time in IHD | 7 days
  Measured using activpal

SECONDARY OUTCOMES:
Posterior wall thickness | 9 months
  Measured in cm
Intraventricular septum | 9 months
  Measured in cm
Left ventricular internal diameter | 9 months
  Measured in cm
Aortic root | 9 months
  Measured in cm
End volume | 9 months
  Measured in cm
E wave | 9 months
  measured in ms
A wave | 9 months
  measured in ms
Relative wall thickness | 9 months
  measured in cm
Left ventricular mass | 9 months
  measured in cm
E/A ratio | 9 months
  ratio between early and late diastolic filling
Isovolumetric relaxation time | 9 months
  measured in ms
Deceleration time | 9 months
  measured in ms
Ejection fraction | 9 months
  presented as a percentage
Stroke volume | 9 months
  measured in litres
Systolic blood pressure | 9 months
  measured in mmHg
Diastolic blood pressure | 9 months
  measured in mmHg
Height | 9 months
  measured in cm
Weight | 9 months
  measured in kg
BMI | 9 months
  measured in kg/m2
Hospital anxiety and depression score | 9 months
  Questions scored out of 3 to determine anxiety and depression level

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT05771610/Prot_000.pdf